CLINICAL TRIAL: NCT00191087
Title: Long-Term Monitoring of Safety in Subjects Treated With Duloxetine for Stress Urinary Incontinence.
Brief Title: Duloxetine in the Treatment of Stress Urinary Incontinence.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2686; F1J-MC-SBAU
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine

SUMMARY:
The purpose of this study is to monitor the long term safety of duloxetine in the treatment of stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Women with predominant stress urinary incontinence.
* 7 or more incontinence episodes per week.

Exclusion Criteria:

* Use of monoamine inhibitors.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458
Dates: Start 2001-04; Study Completion 2006-05

PRIMARY OUTCOMES:
To generate long-term safety data for duloxetine in the treatment of women with stress urinary incontinence

SECONDARY OUTCOMES:
To collect data to demonstrate the maintenance of effect of duloxetine as measured by patient Global Impression of Improvement (PGI-I) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., London, England, United Kingdom